CLINICAL TRIAL: NCT03968614
Title: Electrical Dry Needling as an Adjunct to Eccentric Exercise, Stretching and Manual Therapy for Mid-portion Achilles Tendinopathy: a Multicenter Randomized Clinical Trial
Brief Title: Electrical DN as an Adjunct to Eccentric Exercise, Stretching + MT for Achilles Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, Primary Investigator and President of Spinal Manipulation Institute and Dry Needling Institute of the American Academy of Manipulative Therapy, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT30
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electrical Dry Needling and conventional PT (Experimental): Electrical Dry Needling, Eccentric Exercise, Stretching and Manual Therapy
  Interventions: Other: Electric dry needling and conventional PT
- Conventional PT (Active Comparator): Eccentric Exercise, Stretching and Manual Therapy
  Interventions: Other: Conventional PT

INTERVENTIONS:
Other: Electric dry needling and conventional PT — Electrical Dry Needling, Eccentric Exercise, Stretching and Manual Therapy
  Arms: Electrical Dry Needling and conventional PT
Other: Conventional PT — Eccentric Exercise, Stretching and Manual Therapy
  Arms: Conventional PT

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with achilles tendinopathy: eccentric exercise, stretching and manual therapy VS Electric dry needling, eccentric exercise, stretching and manual therapy. Physical therapists commonly use all of these techniques to treat achilles tendinopathy. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with achilles tendinopathy will be randomized to receive 8-10 treatments (1-2 treatments per week) over 6 weeks (10 treatments max) of either: (1)Eccentric exercise, stretching, manual therapy and electrical dry needling or 2. eccentric exercise, stretching and manual therapy

ELIGIBILITY:
Inclusion Criteria:

1. Adult >18 years old that is able to speak English.
2. Report of at least 3 months of Achilles pain clinically diagnosed as Achilles tendonitis or Achilles tendinopathy
3. Patient has not had physical therapy, massage therapy, chiropractic treatment or injections for Achilles pain in the last 6 months:
4. Diagnosis of noninsertional tendinopathy, defined as the following

   * Subjective report of pain located 2-6 cm proximal to the insertion of Achilles tendon to the calcaneus, particularly with running or jumping
   * Tenderness to palpation of the Achilles tendon while the clinician gently squeezes the tendon between the thumb and index finger in a proximal to distal direction
   * Positive Arc Sign - Intratendinous swelling moves relative to the malleoli with the tendon during active dorsi/plantar Flexion
   * Royal London Test - Tenderness to palpation decreases significantly or disappears with max dorsiflexion

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: hypertension infection, diabetes, peripheral neuropathy, heart disease, stroke, chronic ischemia, edema, severe vascular disease, malignancy, etc.
2. History of previous Achilles tendon surgery, ankle arthrodesis, hind foot fracture, or leg length discrepancy of more than one half inch.
3. History of arthrosis or arthritis of the ankle and/or foot.
4. History of significant ankle and/or foot instability
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   1. Muscle weakness involving a major lower extremity muscle group
   2. Diminished lower extremity patella or Achilles tendon reflexes
   3. Diminished / absent sensation in any lower extremity dermatome
6. Involvement in litigation or worker's compensation regarding foot pain
7. Any condition that might contraindicate the use of electro-needling
8. The patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in VISA-A Questionnaire | baseline, 2 weeks, 6 weeks, 3 months
  Index of severity of Achilles tendinopathy. Lower score means greater severity of condition.

SECONDARY OUTCOMES:
Change in achilles pain (NPRS) (Rating Score) | baseline, 2 weeks, 6 weeks, 3 months
  Higher scores mean greater pain
Change in Foot and Ankle Ability Measure - ADL | baseline, 2 weeks, 6 weeks, 3 months
  activities of daily living (0-84 points) 21 Item 84-point ADL Subscale
Change in Foot and Ankle Ability Measure - Sports | baseline, 2 weeks, 6 weeks, 3 months
  Sports (0-32 points) 8 Item 32-point sports subscale
GROC (ranges from -7 to +7). Global Rating of Change score. | 2 weeks, 6 weeks, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Prisma Health - Research PT Specialists, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No